

## MEDICAL AND HEALTH SCIENCES

## CONSENT FORM THIS FORM WILL BE HELD FOR A PERIOD OF 10 YEARS

Project title: Sustained Wellbeing Benefits of Red Meat Consumption in a Modern Flexitarian Diet: A Study Protocol for a 10 Week Randomised Clinical Trial

Principal Investigator: Dr Andrea Braakhuis (The University of Auckland)

I have read the Participant Information Sheet, have understood the nature of the research and why I have been selected. I have had the opportunity to ask questions and have them answered to my satisfaction. I agree to take part in this research. I have had the opportunity to use support from a family (whānau) member or a fried to help me ask questions and understand the research. I understand that I am free to withdraw participation at any time I understand that blood and saliva samples will be collected and used for research. I understand that samples will be sent around New Zealand and Australia for analysis and disposed of at the end of the study o I wish for a karakia said at the time of my tissue disposal (*please circle*). Yes No I understand that any blood results found to be outside the normal healthy range will be conveyed to me and that if I do not wish to be informed, I cannot participate in this study. I wish to receive the summary of findings. I understand that there may be a No delay between data collection and the publication and availability of the

Name
Signature Date

Researcher's Signature Date

I understand that the results from this study will be used for scientific

I agree not to restrict the use of any data or results that arise from this research

APPROVED BY THE HEALTH AND DISABILITY ETHICS COMMITTEE ON

– 28th January 2021

publication and presentations.

research results (please circle as appropriate).

I wish to receive a copy of my genetic test results

provided such a use is only for scientific purposes.

Reference Number 20/STH/157

Yes

No